CLINICAL TRIAL: NCT00213954
Title: Ultrasound Guidance in Nerve Block Anaesthesia: Classic Nerve Stimulation Technique Versus Ultrasound-Neurostimulation Combination in Four Blocks: Interscalene, Humeral, Parasacral and Lumbar Blocks
Brief Title: Ultrasound Guidance in Nerve Block Anaesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3446; 20050101
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Anesthesia
Keywords: Nerve block anaesthesia; ultrasound-guidance
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- interscalene block (Other): Locoregional anesthesia selection
  Interventions: Procedure: ultrasound-guidance with echography
- axillary block (Other): Locoregional anesthesia selection
  Interventions: Procedure: ultrasound-guidance with echography
- lumbar block (Other): Locoregional anesthesia selection
  Interventions: Procedure: ultrasound-guidance with echography
- parasacral plexus block (Other): Locoregional anesthesia selection
  Interventions: Procedure: ultrasound-guidance with echography

INTERVENTIONS:
Procedure: ultrasound-guidance with echography — Locoregional anesthesia with or without ultrasound guidance practice

SUMMARY:
Nerve block anaesthesia is wildly practised in France, avoiding general anaesthesia in a number of cases and producing excellent post-operative analgesia in trauma and orthopaedic surgeries. Even realised by experimented anaesthetists, 5-15% of failures and rare complications (such as vascular puncture, paresthesia, systemic local anaesthetic toxicity, epidural and spinal anaesthesia, neuropathy) are noticed. The aim of the study is the evaluation of an ultrasound-guidance technique in the four predetermined blocks and the incidence of their complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and greater, scheduled for one of these blocks: interscalene, humeral, parasacral or lumbar blocks, for trauma or orthopaedic surgeries, who have consented to the study and are with social insurance registration

Exclusion Criteria:

* Block's contraindications, treatment by verapamil or flecainide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Estimated)
Dates: Start 2005-05; Primary Completion 2009-03 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Sensory and motor block quality | 15, 30 and 60 min after the block is performed

SECONDARY OUTCOMES:
Complications | during the hospitalisation and by phone 1, 3, 6 and 9 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Laurence LE GOURRIER, MD, Principal Investigator — Unité d'Anesthésiologie et de Réanimation Chirurgicale, Hôpital de Hautepierre
Locations (1):
- Unité d'Anesthésiologie et de Réanimation Chirurgicale, Hôpital de Hautepierre, Strasbourg, France